CLINICAL TRIAL: NCT01556217
Title: A Double-blind, Placebo-controlled, Single Dose, Pharmacokinetic Study to Characterize the Central Brain Penetrance of JNJ-39393406 Using Cerebrospinal Fluid in Healthy Male and Female Subjects
Brief Title: A Pharmacokinetic Study to Characterize JNJ-39393406 in the Cerebrospinal Fluid of Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CR017404; 39393406ALZ1004 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.); 2010-022062-26 (EudraCT Number)
Record Dates: First submitted 2011-04-14; First posted 2012-03-16 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; JNJ-39393406-aaa; Pharmacokinetics; Central brain penetrance; Cerebral spinal fluid
MeSH Terms: interventions — JNJ-39393406

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- JNJ-39393406 (Experimental)
  Interventions: Drug: JNJ-39393406
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-39393406 — Type= exact number, Unit= mg, Number= 200, Form= oral suspension, Route= oral administration. Oral suspension to be taken once with 240 mL (8 ounces of water) between 8:00 AM and 10:30 AM.
  Arms: JNJ-39393406
Drug: Placebo — Form= oral suspension, Route= oral administration. Oral suspension to be taken once with 240 mL (8 ounces of water) between 8:00 AM and 10:30 AM.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the concentration of JNJ-39393406 achieved in the blood and cerebrospinal fluid of healthy adult volunteers following administration of a single dose of JNJ-39393406.

DETAILED DESCRIPTION:
This is a single-centre, double-blind (neither physician nor patient knows the name of the assigned treatment), single dose study of JNJ-39393406 or placebo (a treatment identical in appearance to JNJ-39393406 but does not contain active drug) in healthy adult volunteers. The study consists of an eligibility screening examination (between 21 and 2 days prior to dose administration), a double-blind treatment period, and a follow-up examination (minimally 7 and maximally 14 days after the dose administration). For each volunteer, the maximal study duration will not exceed 6 weeks. JNJ-39393406 or placebo will be administered as a single 200-mg dose on Day 1 as a liquid nanosuspension (a formulation used to improve the solubility of the drug) with 240 mL (approximately 8 ounces or 1 cup) noncarbonated water between 8:00 AM and 10:30 AM after a standard breakfast has been consumed (following a fast [not eating food] of at least 10 hours). Volunteers will then fast until approximately 4 hours after taking JNJ-3939406 or placebo after which lunch will be served.

ELIGIBILITY:
Inclusion Criteria:

* Female volunteers must be postmenopausal (for at least 12 months)
* Body mass index (BMI) between 18 and 29.9 kg/m2, inclusive
* Healthy on the basis of physical examination, neurological examination, medical history, vital signs, and 12-lead ECG [including QTcB interval duration <450 msec] performed at screening. Minor deviations in ECG, which are not considered to be of clinical significance to the investigator, are acceptable
* Healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel [including liver enzymes], hematology, or urinalysis are outside the normal reference ranges, the volunteer may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant

Exclusion Criteria:

* History of liver or renal insufficiency
* significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic disturbances
* Relevant history of or current neurological disease including any history of post dural puncture headache, lower back pain or scoliosis and/or major (lumbar) back surgery, spontaneous, prolonged or severe bleeding with unclear origin, epilepsy or fits or unexplained black-outs
* History or family history of abnormal bleeding or of blood clotting or anemia

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of JNJ39393406 | At 0:30, 1, 1:30, 2, 2:30, 3, 3:30, 4, 6, 8, 10, 12, 16, 20 and 24 hours post dose
Cerebral spinal fluid (CSF) concentration of JNJ39393406 | At 0:30, 1, 1:30, 2, 2:30, 3, 3:30, 4, 6, 8, 10, 12, 16, 20 and 24 hours post dose

SECONDARY OUTCOMES:
Incidence of adverse events as a measure of safety and tolerability | Approximately 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.